CLINICAL TRIAL: NCT03346304
Title: Photodynamic Therapy for the Prevention of Lung Cancer (PEARL)
Brief Title: Photodynamic Therapy for the Prevention of Lung Cancer
Acronym: PEARL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: drug no longer available
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCL/13/0390
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Squamous Cell Lung Cancer; Lung Cancer
Keywords: Autofluorescence Broncoscopy (AFB); Photodynamic Therapy (PDT); High Grade Lesions (HGLs); lung cancer; photosensitiser; Fotolon
MeSH Terms: conditions — Lung Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDT treatment (Intervention Arm) (Experimental): Patients randomised to the PDT treatment (Intervention Arm) will have two courses of PDT treatment in total (for each lung treated). Follow-up is the same as for Control Arm patients: an AFB at 6, 12, 24, and at 36 months post-randomisation; with further AFB visits at 18 and/or at 30 months post-randomisation (dependent on lesion appearance).
  Interventions: Other: Photodynamic Therapy (PDT)
- Surveillance (Control Arm) (No Intervention): Patients randomised to the surveillance (Control Arm) will have: an AFB at 6, 12, 24, and at 36 months post-randomisation; with further AFB visits at 18 and/or at 30 months post-randomisation (dependent on lesion appearance).

INTERVENTIONS:
Other: Photodynamic Therapy (PDT) — Photodynamic Therapy (PDT) using photosensitiser drug Fotolon
  Arms: PDT treatment (Intervention Arm)

SUMMARY:
PEARL is a phase III multicentre 2:1 randomised controlled trial, with an incorporated phase II (pilot) component. All patients consented/registered onto the trial will have an autofluorescence bronchoscopy (AFB) to check for the presence of high grade lesions (HGLs) in the lung, as verified by tissue biopsy. Only patients with one or more histologically confirmed lung HGL will be randomised to receive either photodynamic therapy (PDT) treatment with surveillance (=intervention), or surveillance alone (=control).

The overall aim of the phase II pilot is to demonstrate a >20% response in the PDT group (at least 3 out of 21 PDT patients), compared to a minimum response of 5%. This will be used as an efficacy signal to determine whether the trial will continue into phase III. Response will be measured by regression of high grade lesions (HGLs) to either low grade lesions (LGLs), or to normal epithelium at 6 months post treatment (blind assessment). The overall aim of the phase III is to show that the time period over which HGLs progress to invasive lung cancer is significantly longer when treated with PDT compared to surveillance alone.

DETAILED DESCRIPTION:
Background: Squamous cell carcinoma of the lung develops through a transition of progressive cytological aberration, from normal to metaplasia, mild, moderate, and severe dysplasia and then carcinoma in situ (CIS) before becoming an invasive cancer. Progression rates to invasive carcinoma can vary depending on the initial grade of lesion and it is generally accepted that high-grade lesions are more likely to progress to invasive cancer than low-grade lesions. Early detection and treatment of these lesions is critical to improving survival. There is no evidence base examining how, or whether these high-grade lesions (HGLs) should be treated, resulting in diverse treatment practices both nationally and internationally. This is the first randomised clinical trial of a bronchoscopic intervention in treating HGLs using PDT.

Treatment: Treatment-arm patients will receive two courses of PDT treatment using the photosensitiser drug Fotolon®. Fotolon®, which preferentially accumulates in HGLs, is first administered via IV infusion. Patients then undergo bronchoscopy during which their HGLs are irradiated with red light (via non-heat emitting laser). Red-light activation of the photosensitiser causes chemical transformation of the cells and cell death.

Follow Up: Follow up in both arms consists of AFB surveillance at 6 and 12 months, then every 6-12 months (depending on the appearance of lesions), with annual CT scanning of the thorax, and annual spirometry. Biological samples for translational analysis will be taken at baseline and each subsequent trial visit.

Duration of recruitment: Anticipated recruitment for phase II is 1 year (12 months), and an additional 2 years (24 months) for the phase III.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ≥1 histologically confirmed lung HGL (defined as severe dysplasia or carcinoma in situ) PRE-REGISTRATION: High likelihood of presence of lung HGLs as evaluated by investigator (e.g. because patient part of existing surveillance cohort or referred to trial site) and inclusion/exclusion criteria below. PRE-RANDOMISATION: Following registration and AFB, only patients with ≥1 lung HGLs confirmed histologically can be continue to randomisation provided they continue to meet inclusion/exclusion criteria below.
2. Absence of metastatic disease or other primary cancers as confirmed by CT thorax within 28 days prior to registration only)
3. Male or female patients ≥18 years of age
4. No upper age limit but life expectancy must be at least 3 years
5. ECOG Performance Score 0-2
6. FEV1 ≥ 25% of predicted
7. DLCO/TLCO ≥ 20% of predicted (within 28 days prior to registration only)
8. Women of child-bearing potential (WOCBP), or men with female partners who are pregnant or WOCBP must be willing to practise highly effective methods of birth control starting as soon as possible from the time of informed consent and registration until randomisation (if randomised to the control arm), or until 3 months after the end of their last PDT treatment (if randomised to the intervention arm) . Male patients must also advise their female partners who are WOCBP regarding contraceptive requirements as listed for female patients who are WOCBP.
9. Patients who are WOCBP must also have a negative pregnancy test at the following time points:

   * within 14 days prior to registration
   * within 21 days prior to randomisation
   * and within 24 hours prior to 1st and 2nd PDT treatment, for each lung treated (only if randomised to PDT arm)
10. Ability to give informed consent including the donation of biological samples for translational research

Exclusion criteria:

1. PRE-RANDOMISATION: Finding of (micro)-invasive disease on histology
2. HGLs present for ≥5 years which have remained stable on autofluorescence bronchoscopy (AFB) surveillance
3. Detection of active cancer or on systemic treatment for cancer, excluding basal cell skin cancers (unless adjacent to the illumination site)
4. Previous radiotherapy to the central airways
5. ECOG Performance Score >2
6. Patients who are anticoagulated for prosthetic heart valves
7. Decompensated heart disease with life expectancy less than 3 years
8. Severe liver and renal insufficiency with life expectancy less than 3 years
9. Porphyria or hypersensitivity against porphyrins or photosensitivity
10. Hypersensitivity to chlorine-e6-trisodium salt or therapy with another photosensitising agent or relevant antibiotics (macrolides) in the last 4 weeks
11. Ophthalmic disease likely to require slit-lamp examination within 60 days of registration/randomisation
12. Planned surgical procedure within 60 days of registration/randomisation
13. Patient unlikely to cooperate with a 3-year follow-up; medical or psychological condition at the discretion of the investigator which would not permit compliance with the protocol or meaningful signed informed consent
14. Participation in another study with an investigational medicinal product within one month prior to registration/randomisation
15. Pregnant or breast feeding women (confirmed by serum/urine ß-HCG)
16. Any other condition which is assessed as an intolerable risk by the investigator upon inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Time to site-specific progression | within a 3-year follow-up (incorporates patients from phase II)
  of high grade lesions in the lung to invasive lung cancer; compared between the PDT and control groups

SECONDARY OUTCOMES:
Site-specific response | within a 3-year follow-up (incorporates patients from phase II)
  (regression, stable appearance, progession or recurrence) of HGLs present at baseline (index lesions); compared between the PDT and control groups
Number of new HGLs | within a 3-year follow-up (incorporates patients from phase II)
  HGLs identified post-baseline at new sites within the lung (i.e. not at the site of the index lesions); compared between the PDT and control groups
Number of metachronous endobronchial lung cancers | within a 3-year follow-up (incorporates patients from phase II)
  that develop at remote sites within the lung in both arms
Cumulative risk of developing lung cancer | within a 3-year follow-up (incorporates patients from phase II)
  as detected on bronchoscopy and CT thorax in patients harbouring HGLs from date of randomisation; compared between the PDT and control groups
Overall and cancer specific survival | within a 3-year follow-up (incorporates patients from phase II)
  from date of randomisation; compared between the PDT and control groups
Difference in spirometry (FEV1, FVC) values | at specific time points (6,12,24 and 36 months post randomisation);
  to determine whether PDT affects spirometry
Adverse events | within a 3-year follow-up (incorporates patients from phase II)
  Based on the maximum toxicity grade for each patient for each event type; compared between the PDT and control groups
EQ-5D-5L | at specific time points (6,12,24 and 36 months, and possibly 18 and 30 months, post randomisation); compared between the PDT and control groups
  Health-Related Quality of Life (HRQoL)
EORTC QLQ-LC13 | at specific time points (6,12,24 and 36 months, and possibly 18 and 30 months, post randomisation); compared between the PDT and control groups
  Health-Related Quality of Life (HRQoL)
ACE-27 | at specific time points (6,12,24 and 36 months, and possibly 18 and 30 months, post randomisation); compared between the PDT and control groups
  Health-Related Quality of Life (HRQoL)

IPD SHARING:
Plan to Share IPD: No